CLINICAL TRIAL: NCT01222117
Title: A Phase 2, Randomized, Open-label (With Blinded Plasminogen Activator and Placebo Control Groups) Study to Evaluate the Effects of Different Intra-thrombus Infusion Regimens of Plasmin (Human) Compared to Plasminogen Activator and Placebo In Patients With Acute Lower Extremity Native Artery or Bypass Graft Occlusion
Brief Title: A Study of Intra-thrombus Plasmin (Human) In Acute Peripheral Arterial Occlusion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T05018-2004; 2010-019760-36 (EudraCT Number)
Record Dates: First submitted 2010-10-13; First posted 2010-10-18 (Estimated); Results first posted 2016-05-30 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2016-11

CONDITIONS: Acute Peripheral Arterial Occlusion
Keywords: Acute Limb Ischemia
MeSH Terms: interventions — Fibrinolysin; Plasminogen Activators; Tissue Plasminogen Activator; Urokinase-Type Plasminogen Activator; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (11):
- Plasmin Open-label Treatment Group A (Experimental): Open-label 150 mg Plasmin administered without initial proximal pulse; 5-hour infusion using 10 mL/hour infusion rate.
  Interventions: Biological: Plasmin
- Plasmin Open-label Treatment Group B (Experimental): Open-label 150 mg Plasmin administered with initial proximal pulse; 5-hour infusion using 15 mL/hour infusion rate
  Interventions: Biological: Plasmin
- Plasmin Open-label Treatment Group C (Experimental): Open-label 150 mg Plasmin administered with proximal pulse; 5 hour infusion using 30 mL/hour infusion rate.
  Interventions: Biological: Plasmin
- Plasmin Open-label Treatment Group D (Experimental): Open-label 150 mg Plasmin administered with proximal pulse; 2-hour infusion using 35 mL/hour infusion rate
  Interventions: Biological: Plasmin
- Plasminogen Activator Blinded Group E (Active Comparator): PA administered for five hours at a dose and volume according to the Investigator's clinical judgement/standard practice
  Interventions: Biological: Plasminogen Activator
- PA Placebo Blinded Treatment Arm F (Placebo Comparator): PA placebo (normal saline for injection) administered for five hours at a dose and volume according to the Investigator's clinical judgement/standard practice for PA administration
  Interventions: Other: Placebo
- Plasmin Open-label Treatment Group G (Experimental): Open-label 150 mg Plasmin administered without pulsing; 5-hour infusion using 60 mL/hour infusion rate
  Interventions: Biological: Plasmin
- Plasmin Open-label Treatment Group H (Experimental): Open-label 150 mg Plasmin administered without pulsing; 2-hour infusion using 75 mL/hour infusion rate
  Interventions: Biological: Plasmin
- Plasmin Open-label Treatment Group I (Experimental): Open-label 150 mg Plasmin administered without pulsing; 5-hour infusion using 30 mL/hour infusion rate with balloon occlusion catheter
  Interventions: Biological: Plasmin
- Plasmin Open-label Treatment Group J (Experimental): Open-label 150 mg Plasmin administered without pulsing; 2-hour infusion using 35 mL/hour infusion rate with balloon occlusion catheter
  Interventions: Biological: Plasmin
- Plasmin Open-label Treatment Group M (Experimental): Open-label 250 mg Plasmin administered without pulsing; 5-hour infusion using 30 mL/hour infusion rate with balloon occlusion catheter
  Interventions: Biological: Plasmin

INTERVENTIONS:
Biological: Plasmin — Plasmin prepared in 0.9% saline for injection
  Other Names: Plasmin (Human)
  Arms: Plasmin Open-label Treatment Group A; Plasmin Open-label Treatment Group B; Plasmin Open-label Treatment Group C; Plasmin Open-label Treatment Group D; Plasmin Open-label Treatment Group G; Plasmin Open-label Treatment Group H; Plasmin Open-label Treatment Group I; Plasmin Open-label Treatment Group J; Plasmin Open-label Treatment Group M
Biological: Plasminogen Activator — Plasminogen activator used according to the Investigator's clinical judgment.
  Other Names: tissue plasminogen activator (tPA); urokinase (UK)
  Arms: Plasminogen Activator Blinded Group E
Other: Placebo — Normal saline for injection at the same volume as the plasminogen activator.
  Other Names: Normal saline
  Arms: PA Placebo Blinded Treatment Arm F

SUMMARY:
The primary purpose of this Phase 2 study is to optimize Plasmin delivery by comparing different delivery regimens in patients with peripheral arterial occlusion. The study includes a blinded plasminogen activator treatment group and a blinded plasminogen activator placebo group. The study will also assess safety and tolerability of Plasmin at 150 and 250 mg doses.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral limb ischemia - Society of Vascular Surgery Categories I and IIa
* Onset of symptoms less than or equal to 14 days
* Thrombosed infrainguinal bypass graft or native artery
* Diagnosis by arteriography of occlusive thrombus in graft or artery
* Ability to embed the infusion catheter into the thrombus
* Women of childbearing potential must use contraception and have a negative pregnancy test

Exclusion Criteria:

* Any medical or social condition that may interfere with study participation
* Women who are pregnant or lactating
* Hemorrhagic stroke history
* Thrombotic or embolic stroke or cerebrovascular events (including transient ischemic attack) within one year
* Intracranial or spinal neurosurgery, or severe intracranial trauma in the last 3 months
* Major surgery, organ biopsy, or major trauma within the past 10 days
* Lumbar puncture or non-compressible arterial puncture in the past 10 days
* Intraocular surgery within the past 10 days
* Active gastrointestinal or organ bleeding
* Uncontrolled arterial hypertension (systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg)
* Known intracranial neoplasm, aneurysm, or arteriovenous malformation
* Current bleeding diathesis
* Platelet count <75 x 10e9/L
* Active graft infection
* Occlusion occurred within one month of synthetic graft placement
* Occlusion occurred within 6 months of autologous graft placement
* A sequential composite graft with dual outflows to correct multiple occlusions
* Medically unable to tolerate an open vascular procedure
* Known prothrombotic state
* Hemoglobin <10.0 g/dL
* Impaired renal function or renal disease that constitutes a contraindication to contrast angiography, including creatinine >2.0 mg/dL
* Treatment with a full dose plasminogen activator (PA) within the last 48 hours
* Treatment with a glycoprotein IIb/IIIa class of platelet inhibitor within the past 5 days
* Treatment with oral anticoagulants, and with an international normalized ratio of >1.7

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2010-12; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kecia Courtney, Study Director — Grifols Therapeutics
Locations (39):
- United States (2):
  - Kaleida Health System, Buffalo, New York
  - Cleveland Clinic, Cleveland, Ohio
- Belgium (4):
  - Ziekenhuis Oost Limburg, Campus St. Jan, Genk, Limburg
  - Erasme Hospital, Brussels, Brussels
  - University Hospital Antwerp, Edegem
  - Chirurgie UZ Leuven, Leuven
- Bulgaria (2):
  - Clinic of Vascular Surgery and Angiology, Sofia
  - Tokuda Hospital Sofia, Sofia
- Czechia (5):
  - Vascular Centre Vitkovicka Nemocnice, Ostrava - Vitkovice
  - Cevni Chirurgie, Nemocnice Na Homolce, Prague
  - IKEM, Kardiologicka klinika, Prague
  - University Hospital Kralovske Vinobrady, Prague
  - Chirurgicka klinika IPVZ, Ústí nad Labem
- Germany (3):
  - Universitätsklinikum Bonn, Radiologische Universitätsklinik, Bonn
  - Universitäts GefäßCentrum Uniklinikum Dresden, Dresden
  - Klinik für Innere Medizin I - Angiologie / Kardiologie, Leipzig
- India (2):
  - Life Care Institute of Medical Sciences and Research, Gujarat
  - Gokula Metropolis Clinical Research Centre, M. S. Ramaiah Hospital, Karnataka
- Peru (4):
  - Centro de Investigación y Atención Cardiovascular, Lima
  - Hospital Nacional Edgardo Rebagliati Martins, Lima
  - Hospital Nacional Guillermo Almenara Irigoyen-EsSalud, Lima
  - Instituto Neuro Cardiovascular de las Americas, Lima
- Poland (6):
  - Wojewodzki Szpital Specjalistyczny nr 4 w Bytomiu, Bytom
  - Malopolskie Centrum Sercowo-Naczyniowe PAKS American Heart of Poland Sp. z o.o, Chrzanów
  - Uniwersyleckie Centrum Kliniczne, Gdansk
  - Szpital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Poznan
  - Zaklad Opieki Zdrowonej Ministerstwa Spraw Wewnetrznych i Administracji w Poznaniu, Poznan
  - Samodzielny Publiczny Szpital Kliniczny Nr 2 PUM w Szczecinie, Szczecin
- Romania (4):
  - Institutul de Urgenta pentru Boli Cardiovasculare "Prof.Dr.C.C.Iliescu", Bucharest
  - Institutul Inimii "Nicolae Stancioiu" Cluj-Napoca, Cluj-Napoca
  - Inst.de Boli Cardiovasculare "Prof.I.M.Georgescu" Iasi, Iași
  - Institutul de Boli Cardiovasculare si Transplant Mures, Târgu Mureş
- Serbia (4):
  - Institut za kardiovaskularne bolesti Dedinje, Belgrade
  - Klinicki Centar Srbije, Belgrade
  - Klinicki Centar Nis, Niš
  - Klinicki Centar Vojvodine, Novi Sad
- Slovakia (2):
  - Oddelenie diagnostickej a intervencnej radiologie, The National Institute of Cardiovascular Diseases, Bratislava
  - The Eastern Slovak Institute of Cardiovascular Diseases, Košice
- Fundacion Hospital Alcorcon, Alcorcón, Spain

REFERENCES:
- [Derived] Comerota AJ, Davidovic L, Hanna K, Courtney KL, Shlansky-Goldberg RD. Phase 2, randomized, open-label study on catheter-directed thrombolysis with plasmin versus rtPA and placebo in acute peripheral arterial occlusion. J Drug Assess. 2019 Apr 9;8(1):43-54. doi: 10.1080/21556660.2019.1586402. eCollection 2019. PMID 31069128

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Plasmin Open-label Treatment Group A | Plasmin Open-label Treatment Group B | Plasmin Open-label Treatment Group C | Plasmin Open-label Treatment Group D | Plasminogen Activator Blinded Group E | PA Placebo Blinded Treatment Arm F | Plasmin Open-label Treatment Group G | Plasmin Open-label Treatment Group H | Plasmin Open-label Treatment Group I | Plasmin Open-label Treatment Group J | Plasmin Open-label Treatment Group M
Started | 20 | 20 | 22 | 20 | 9 | 10 | 13 | 12 | 23 | 19 | 6
Completed | 17 | 19 | 22 | 19 | 8 | 9 | 13 | 12 | 20 | 17 | 6
Not Completed | 3 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 3 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Plasminogen Activator Blinded Group E: PA administered for 5 hours at a dose and volume according to the Investigator's clinical judgement/standard practice
  Plasminogen Activator: Plasminogen activator used according to the Investigator's clinical judgment.
- PA Placebo Blinded Treatment Arm F: PA placebo (normal saline for injection) administered for 5 hours at a dose and volume according to the Investigator's clinical judgement/standard practice for PA administration
  Placebo: Normal saline for injection at the same volume as the plasminogen activator.
- Total: Total of all reporting groups
Arm/Group | Plasmin Open-label Treatment Group A | Plasmin Open-label Treatment Group B | Plasmin Open-label Treatment Group C | Plasmin Open-label Treatment Group D | Plasminogen Activator Blinded Group E | PA Placebo Blinded Treatment Arm F | Plasmin Open-label Treatment Group G | Plasmin Open-label Treatment Group H | Plasmin Open-label Treatment Group I | Plasmin Open-label Treatment Group J | Plasmin Open-label Treatment Group M | Total
Number analyzed (Participants) | 20 | 20 | 22 | 20 | 9 | 10 | 13 | 12 | 23 | 19 | 6 | 174
Age, Customized [Number; unit: participants]
  <65 years | 12 | 10 | 10 | 10 | 5 | 5 | 8 | 7 | 13 | 12 | 3 | 95
  >=65 years | 8 | 10 | 12 | 10 | 4 | 5 | 5 | 5 | 10 | 7 | 3 | 79
Gender [Count of Participants; unit: Participants]
  Female | 3 | 3 | 5 | 7 | 0 | 3 | 2 | 3 | 7 | 5 | 1 | 39
  Male | 17 | 17 | 17 | 13 | 9 | 7 | 11 | 9 | 16 | 14 | 5 | 135
Region of Enrollment [Number; unit: participants]
  Czech Republic | 4 | 4 | 3 | 5 | 1 | 1 | 5 | 5 | 9 | 7 | 1 | 45
  Romania | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Belgium | 3 | 1 | 3 | 2 | 2 | 2 | 1 | 0 | 1 | 0 | 0 | 15
  United States | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5
  Poland | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 5
  Slovakia | 3 | 2 | 4 | 1 | 1 | 0 | 2 | 2 | 11 | 9 | 5 | 40
  Serbia | 6 | 7 | 3 | 4 | 4 | 6 | 4 | 5 | 1 | 3 | 0 | 43
  Bulgaria | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5
  Peru | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Germany | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  India | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Ukraine | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects With >50% Thrombolysis
Description: The proportion of subjects with >50% thrombolysis at the end of treatment compared to baseline by arteriography.
Time Frame: 5 hours (Treatment Groups A, B, C, G, I, M) or 2 hours (Treatment Groups D, H, J)
Population: In groups A-D, G and H, 8 subjects were excluded (EOT arteriogram missing or not read, did not receive >=90% of dose). In groups I and J, 11 subjects were excluded (BOC not inserted/appropriately inflated, missing an arteriogram). In group F, 1 subject was not dosed and 4 subjects were excluded (did not receive >=90% of dose).
Measure: Number; unit: percentage of participants
Arm/Group | Plasmin Open-label Treatment Group A | Plasmin Open-label Treatment Group B | Plasmin Open-label Treatment Group C | Plasmin Open-label Treatment Group D | Plasminogen Activator Blinded Group E | PA Placebo Blinded Treatment Arm F | Plasmin Open-label Treatment Group G | Plasmin Open-label Treatment Group H | Plasmin Open-label Treatment Group I | Plasmin Open-label Treatment Group J | Plasmin Open-label Treatment Group M
Number analyzed (Participants) | 16 | 19 | 21 | 19 | 9 | 5 | 12 | 12 | 15 | 14 | 6
percentage of participants | 43.8 | 47.4 | 81.0 | 47.4 | 88.9 | 40.0 | 66.7 | 66.7 | 73.3 | 42.9 | 33.3

2. Secondary Outcome: The Incidence of Major and Minor Bleeding Events, Deaths, Adverse Events, Serious Adverse Events, and Abnormal Laboratory Values as a Measure of Safety and Tolerability.
Description: The incidence of major and minor bleeding events, deaths, adverse events, serious adverse events, and abnormal laboratory values as a measure of safety and tolerability.
Time Frame: 30 days
Population: Subjects were excluded from the safety population if they did not receive any dose of Plasmin (groups I and J) or placebo (group F)
Measure: Number; unit: percentage of participants
Arm/Group | Plasmin Open-label Treatment Group A | Plasmin Open-label Treatment Group B | Plasmin Open-label Treatment Group C | Plasmin Open-label Treatment Group D | Plasminogen Activator Blinded Group E | PA Placebo Blinded Treatment Arm F | Plasmin Open-label Treatment Group G | Plasmin Open-label Treatment Group H | Plasmin Open-label Treatment Group I | Plasmin Open-label Treatment Group J | Plasmin Open-label Treatment Group M
Number analyzed (Participants) | 20 | 20 | 22 | 20 | 9 | 9 | 13 | 12 | 21 | 17 | 6
percentage of participants
  Adverse events | 80.0 | 60.0 | 81.8 | 70.0 | 77.8 | 88.9 | 69.2 | 58.3 | 66.7 | 58.8 | 50.0
  Serious adverse events | 50.0 | 20.0 | 27.3 | 20.0 | 22.2 | 55.6 | 30.8 | 25.0 | 33.3 | 11.8 | 0
  Major bleeding events | 15.0 | 5.0 | 4.5 | 0 | 11.1 | 11.1 | 0 | 0 | 9.5 | 0 | 0
  Minor bleeding events | 5.0 | 20.0 | 9.1 | 20.0 | 33.3 | 33.3 | 46.2 | 8.3 | 28.6 | 11.8 | 33.3
  Deaths | 5.0 | 0 | 0 | 0 | 11.1 | 11.1 | 0 | 0 | 0 | 0 | 0
  Abnormal laboratory values | 15.0 | 10.0 | 13.7 | 0 | 11.1 | 22.2 | 15.4 | 0 | 4.8 | 0 | 0

ADVERSE EVENTS:
Description: Subjects were excluded from the safety population if they did not receive any dose of Plasmin (groups I and J) or placebo (group F)
Arm/Group | Plasmin Open-label Treatment Group A | Plasmin Open-label Treatment Group B | Plasmin Open-label Treatment Group C | Plasmin Open-label Treatment Group D | Plasminogen Activator Blinded Group E | PA Placebo Blinded Treatment Arm F | Plasmin Open-label Treatment Group G | Plasmin Open-label Treatment Group H | Plasmin Open-label Treatment Group I | Plasmin Open-label Treatment Group J | Plasmin Open-label Treatment Group M
Serious Adverse Events (participants affected / at risk) | 10/20 | 4/20 | 6/22 | 4/20 | 2/9 | 5/9 | 4/13 | 3/12 | 7/21 | 2/17 | 0/6
Other Adverse Events (participants affected / at risk) | 14/20 | 11/20 | 18/22 | 14/20 | 7/9 | 8/9 | 7/13 | 5/12 | 12/21 | 10/17 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Plasmin Open-label Treatment Group A (N=20) | Plasmin Open-label Treatment Group B (N=20) | Plasmin Open-label Treatment Group C (N=22) | Plasmin Open-label Treatment Group D (N=20) | Plasminogen Activator Blinded Group E (N=9) | PA Placebo Blinded Treatment Arm F (N=9) | Plasmin Open-label Treatment Group G (N=13) | Plasmin Open-label Treatment Group H (N=12) | Plasmin Open-label Treatment Group I (N=21) | Plasmin Open-label Treatment Group J (N=17) | Plasmin Open-label Treatment Group M (N=6)
Peripheral ischaemia (Vascular disorders) | 4 | 0 | 1 | 2 | 0 | 3 | 0 | 2 | 0 | 0 | 0
Peripheral embolism (Vascular disorders) | 4 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Reocclusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Ischaemia (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femoral arterial stenosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Graft thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arterial thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Ischaemic limb pain (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Reperfusion injury (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Puncture site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Plasmin Open-label Treatment Group A (N=20) | Plasmin Open-label Treatment Group B (N=20) | Plasmin Open-label Treatment Group C (N=22) | Plasmin Open-label Treatment Group D (N=20) | Plasminogen Activator Blinded Group E (N=9) | PA Placebo Blinded Treatment Arm F (N=9) | Plasmin Open-label Treatment Group G (N=13) | Plasmin Open-label Treatment Group H (N=12) | Plasmin Open-label Treatment Group I (N=21) | Plasmin Open-label Treatment Group J (N=17) | Plasmin Open-label Treatment Group M (N=6)
Peripheral embolism (Vascular disorders) | 4 | 2 | 6 | 1 | 1 | 1 | 2 | 0 | 4 | 3 | 0
Haematoma (Vascular disorders) | 0 | 2 | 1 | 2 | 3 | 1 | 4 | 1 | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arterial thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 2
Hypertension (Vascular disorders) | 1 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Femoral artery embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic limb pain (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Extremity necrosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Iliac artery stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Labile blood pressure (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral artery dissection (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion related reaction (General disorders) | 5 | 2 | 5 | 6 | 2 | 4 | 0 | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 0 | 1 | 3 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Puncture site haemorrhage (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Oedema peripheral (General disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion site haemorrhage (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Reocclusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematocrit decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Hypercoagulation (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Graft infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Device leakage (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Red blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vascular graft complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Complication of device removal (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site haematoma (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood fibrinogen decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Postoperatvie wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral artery aneurysm (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the study, after providing sponsor 30 days' notice prior to submitting a manuscript or other materials related to the study to any outside party. At sponsor's request, site will remove any confidential information (other than study results), and site will upon sponsor's request delay publication or presentation for a period of up to 60 days to allow sponsor to protect its interests in any sponsor inventions